CLINICAL TRIAL: NCT00185107
Title: A Multi-Center, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study of the Efficacy and Safety of WelChol® in Combination With Zetia® Compared to Zetia® Alone in Patients With Primary Hypercholesterolemia
Brief Title: Effect of Combination Therapy With Two Drugs (Colesevelam and Ezetimibe) in Patients With High Cholesterol
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WEL-408
Record Dates: First submitted 2005-09-09; First posted 2005-09-16 (Estimated); Last update posted 2007-09-11 (Estimated); Status verified 2007-09

CONDITIONS: Hypercholesterolemia
Keywords: Safety; Efficacy; WelChol®; Zocor®; Zetia®
MeSH Terms: conditions — Hypercholesterolemia | interventions — Colesevelam Hydrochloride; Ezetimibe; Simvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Colesevelam Hydrochloride
Drug: Ezetimibe
Drug: Simvastatin

SUMMARY:
Assess the efficacy of WelChol® plus Zetia® in treating patients with high cholesterol

ELIGIBILITY:
Inclusion Criteria:

* 18-80 years of age, inclusive;
* A history of primary hypercholesterolemia

Exclusion Criteria:

* Any serious disorders including pulmonary, hepatic, renal, gastrointestinal (including clinically significant malabsorption), uncontrolled endocrine/ metabolic, hematologic/oncologic (within the last 5 years), neurologic and psychiatric diseases that would interfere with the conduct of the study or interpretation of the data;
* Hepatic dysfunction including biliary cirrhosis, unexplained persistent liver function abnormality, and pre-existing gallbladder disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45
Dates: Start 2005-03; Study Completion 2005-10

PRIMARY OUTCOMES:
The percent change in LDL-C from the start of the study

SECONDARY OUTCOMES:
- The absolute change in LDL-C from baseline
- The percent change in LDL-C from baseline
- The absolute changes and percent changes in TG, non-HDL-
C, HDL-C, total cholesterol and other lipid measures
- The percentages of patients who achieve target levels of LDL-C at the end of the study

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Scripps Clinic, San Diego, California
  - Renstar Medical Research, Ocala, Florida
  - Radiant Research, Overland Park, Kansas
  - L-MARC Research Center, Louisville, Kentucky
  - Radiant Research, Edina, Minnesota
  - Medical Office, Statesville, North Carolina
  - Linder Clinical Trial Center, Cincinnati, Ohio